CLINICAL TRIAL: NCT02170727
Title: A Phase 3 Study of a Daclatasvir/Asunaprevir/BMS-791325 Fixed Dose Combination (FDC) in Subjects With Chronic Hepatitis C Genotype 1
Acronym: UNITY 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI443-123
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 : DCV/ASV/BMS-791325 (Experimental): DCV 30 mg (as the free base) / Asunaprevir (ASV) 200 mg / BMS-791325 75 mg FDC tablet orally twice daily for 12 weeks
  Interventions: Drug: DCV/ASV/BMS-791325

INTERVENTIONS:
Drug: DCV/ASV/BMS-791325

SUMMARY:
To demonstrate the effectiveness of Daclatasvir (DCV) 3 Direct Acting Antivirals (DAA) fixed dose combination in Genotype 1 Chronic Hepatitis C subjects.

DETAILED DESCRIPTION:
US National Institutes of Health Division of AIDs (DAIDS)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subject chronically infected with HCV genotype 1 (GT-1)
* Subject without cirrhosis or with compensated cirrhosis (Child Pugh Class A)
* HCV RNA ≥ 10,000 IU/mL at screening
* Treatment-naïve subject with no previous exposure to an interferon formulation (ie, IFNα, pegIFNα), Ribavirin (RBV), or HCV DAA (protease, polymerase inhibitor, etc.)
* Interferon (IFN) experienced subject who have received previous treatment with IFNα, with or without RBV

Exclusion Criteria:

* Liver or any other transplant (including hematopoietic stem cell transplants) other than cornea and hair;
* Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to screening;
* Documented or suspected hepatocellular carcinoma (HCC), as evidenced by previously obtained imaging studies or liver biopsy (or on a screening imaging study/liver biopsy if this was performed);
* Evidence of decompensated liver disease including, but not limited to, radiologic criteria, a history or presence of ascites, bleeding varices, or hepatic encephalopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2015-06-12 (Actual); Study Completion 2015-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- Russia (2):
  - Local Institution, Kazan'
  - Local Institution, Moscow
- South Korea (5):
  - Local Institution, Busan
  - Local Institution, Gyeonggi-do
  - Local Institution, Gyeongsangnam-do
  - Local Institution, Inchoen
  - Local Institution, Seoul
- Taiwan (5):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
  - Local Institution, Taoyuan District

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 169 subjects were treated; 138 treatment-naive and 31 treatment-experienced; 3 participants did not complete the treatment period (1 was lost to follow-up and 2 had withdrawn)
Groups:
- Treatment-Naive: DCV/ASV/BMS-791325: Daclatasvir (DCV) 30 mg/ Asunaprevir (ASV) 200 mg / BMS-791325 75 mg FDC tablet orally twice daily for 12 weeks
- Treatment-Experianced:: Daclatasvir (DCV) 30 mg / Asunaprevir (ASV) 200 mg / BMS-791325 75 mg FDC tablet orally twice daily for 12 weeks
Period: Overall Study
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
Started | 138 | 31
Completed | 135 | 31
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced: | Total
Number analyzed (Participants) | 138 | 31 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.78) | 53.0 (12.64) | 52.2 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 11 | 81
  Male | 68 | 20 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 128 | 31 | 159
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 0 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Asia | 128 | 31 | 159
  Europe | 10 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 (SVR12) in the Naive Cohort
Description: Percentage of Participants with SVR12 in the naive cohort, defined as HCV RNA < LLOQ target detected (TD) or target not detected (TND) (LOQ TD/TND) at post-treatment follow-up Week 12.
Time Frame: Post treatment Week 12
Population: Analysis population included enrolled participants who received at least 1 dose of study therapy. SVR12 was based on Next Value Carried Backwards approach. (Exact binomial confidence interval reported)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325
Number analyzed (Participants) | 138
Percentage of Participants | 98.6 [94.9 to 99.8]

2. Secondary Outcome: Percentage of Participants With SVR12 in the Interferon Alfa (IFN-a) Experienced Cohort
Description: Percentage of treated participants with SVR12 in the IFNα experienced cohort, defined as HCV RNA < LLOQ target detected or target not detected (LLOQ TD/TND).
Time Frame: Post treatment Week 12
Population: Analysis population included enrolled participants who received at least 1 dose of study therapy. SVR12 was based on Next Value Carried Backwards approach.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325
Number analyzed (Participants) | 31
Percentage of Participants | 100.0 [88.8 to 100.0]

3. Secondary Outcome: Percentage of Participants Who Achieved HCV RNA < LLOQ TD/TND
Description: Percentage of Participants with hepatitis C virus(HCV) ribonucleic acid (RNA) < lower limit of quantitation (LLOQ), target detected (TD) or target not detected (TND) were presented at treatment Weeks 1, 2, 4, 6, 8, 12, EOT, and follow-up Weeks 4 (SVR4), 8 (SVR8), and 24 (SVR24).
Time Frame: On-treatment Weeks: 1, 2, 4, 6, 8, and 12; post treatment Weeks 4 (SVR4), 8 (SVR8), 24 (SVR24) and EOT (end of treatment)
Population: Included participants who received 1 dose of study therapy. SVR24 based on Observed Values approach. Participants with missing HCV RNA results at follow-up Week 24 were considered non-responders for SVR24. SVR12 is based on Next Value Carried Backwards approach and modified ITT (intent-to-treat) analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
Number analyzed (Participants) | 138 | 31
Percentage of Participants
  Week 1 | 44.2 [35.9 to 52.5] | 29.0 [14.2 to 48.0]
  Week 2 | 87.7 [82.2 to 93.2] | 80.6 [62.5 to 92.5]
  Week 4 | 99.3 [96.0 to 100.0] | 93.5 [78.6 to 99.2]
  Week 6 | 100.0 [97.4 to 100.0] | 100.0 [88.8 to 100.0]
  Week 8 | 99.3 [96.0 to 100.0] | 100.0 [88.8 to 100.0]
  Week 12 | 100.0 [97.4 to 100.0] | 96.8 [83.3 to 99.9]
  End of Treatment | 100.0 [97.4 to 100.0] | 100.0 [88.8 to 100.0]
  Follow-Up Week 4 | 97.8 [93.8 to 99.5] | 96.8 [83.3 to 99.9]
  Follow-Up Week 8 | 98.6 [94.9 to 99.8] | 96.8 [83.3 to 99.9]
  Follow-Up Week 24 | 96.4 [91.7 to 98.8] | 100.0 [88.8 to 100.0]

4. Secondary Outcome: Percentage of Participants Who Achieved HCV RNA < LLOQ TND
Description: Percentage of treated participants with HCV RNA < LLOQ, TND (target not detected) were presented at treatment Weeks 1, 2, 4, 6, 8, 12, at both Weeks 4 and 12, EOT, and follow-up Weeks 4, 8, 12 and 24.
Time Frame: On-treatment Weeks: 1, 2, 4, 6, 8, and 12 and post treatment weeks 4, 8, 12, 24 and EOT (end of treatment)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
Number analyzed (Participants) | 138 | 31
Percentage of Participants
  Week 1 | 11.6 [6.3 to 16.9] | 0.0 [0.0 to 11.2]
  Week 2 | 42.0 [33.8 to 50.3] | 25.8 [11.9 to 44.6]
  Week 4 | 93.5 [89.4 to 97.6] | 90.3 [74.2 to 98.0]
  Week 6 | 98.6 [94.9 to 99.8] | 100.0 [88.8 to 100.0]
  Week 8 | 99.3 [96.0 to 100.0] | 100.0 [88.8 to 100.0]
  Week 12 | 97.8 [93.8 to 99.5] | 96.8 [83.3 to 99.9]
  End of Treatment | 97.8 [93.8 to 99.5] | 100.0 [88.8 to 100.0]
  Follow-Up Week 4 | 97.1 [92.7 to 99.2] | 96.8 [83.3 to 99.9]
  Follow-Up Week 8 | 98.6 [94.9 to 99.8] | 96.8 [83.3 to 99.9]
  Follow-Up Week 12 | 98.6 [94.9 to 99.8] | 100.0 [88.8 to 100.0]
  Follow-Up Week 24 | 96.4 [91.7 to 98.8] | 100.0 [88.8 to 100.0]

5. Secondary Outcome: Number of Participants With Deaths, Serious Adverse Events (SAEs) and AEs Leading to Discontinuation From Treatment
Description: SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/ birth defect.
Time Frame: Up to post treatment week 4
Population: Safety analysis population included participants who received at least 1 dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
Number analyzed (Participants) | 138 | 31
Participants
  Serious Adverse Events | 2 | 0
  AEs Leading to Discontinuation | 2 | 2
  Deaths | 0 | 0

6. Secondary Outcome: Percentage of Participants With Anemia Defined as Hb < 10 g/dL On-treatment Who Had Hb >=10 g/dL at Baseline
Description: Anemia was defined as hemoglobin < 10 g/dL on-treatment for subjects who had hemoglobin >= 10 g/dL at baseline.
Time Frame: Up to post treatment week 4
Population: Analysis population included enrolled participants who received at least 1 dose of study therapy
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
Number analyzed (Participants) | 138 | 31
Percentage of Participants | 1.4 [0.0 to 3.4] | 0.0 [0.0 to 0.0]

7. Secondary Outcome: Percentage of Participants Who Achieved SVR12 Associated With Hepatitis C Virus (HCV) Genotype Subtype 1a vs 1b
Description: Percentage of subjects in each cohort who achieved SVR12 associated with HCV genotype subtype 1a vs 1b were reported.
Time Frame: Post treatment week 12
Population: It included enrolled participants who received at least 1 dose of study therapy. Here, N signifies number of participants evaluable for the outcome measure, 'n' signifies number of participants analysed for specific category. SVR12 is based on Next Value Carried Backwards approach
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
Number analyzed (Participants) | 136 | 31
Percentage of participants
  Genotype - 1a: number analyzed (Participants) | 9 | 2
  Genotype - 1a | 88.9 [51.8 to 99.7] | 100.0 [15.8 to 100.0]
  Genotype - 1b: number analyzed (Participants) | 128 | 29
  Genotype - 1b | 100.0 [97.2 to 100.0] | 100.0 [88.1 to 100.0]

8. Secondary Outcome: Proportion of Participants Who Achieved SVR12 Associated With IL28B rs12979860 Single Nucleotide Polymorphisms (SNP) Status (CC Genotype or Non CC Genotype)
Description: Proportion of Participants who Achieved SVR12 Associated with IL28B rs12979860 Single Nucleotide Polymorphisms (SNP) status (CC genotype or non CC genotype) were reported.
Time Frame: Post treatment Week 12
Population: It included enrolled participants who received at least 1 dose of study therapy. SVR12 is based on Next Value Carried Backwards approach
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
Number analyzed (Participants) | 138 | 31
Percentage of Participants
  CC genotype: number analyzed (Participants) | 98 | 18
  CC genotype | 99.0 | 100.0
  Non-CC Genotype: number analyzed (Participants) | 39 | 13
  Non-CC Genotype | 97.4 | 100.0

9. Secondary Outcome: Proportion of Cirrhotic and Non Cirrhotic Participants Who Achieved SVR12
Description: Proportion of Cirrhotic and Non Cirrhotic Participants who Achieved SVR12 were reported.
Time Frame: Post treatment Week 12
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
Number analyzed (Participants) | 138 | 31
Percentage of Participants
  Cirrhotic: number analyzed (Participants) | 16 | 7
  Cirrhotic | 100.0 | 100.0
  Noncirrhotic: number analyzed (Participants) | 122 | 24
  Noncirrhotic | 98.4 | 100.0

10. Secondary Outcome: Number of Participants With Selected Grade 3/4 Laboratory Abnormalities
Description: Rates of selected Grade 3 - 4 laboratory abnormalities on treatment in each cohort was estimated
Time Frame: Post treatment week 4
Population: Safety analysis population included participants who received at least 1 dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
Number analyzed (Participants) | 138 | 31
Participants | 16 | 5

11. Secondary Outcome: Number of Participants With/Without Cirrhosis as Measured by SAEs and Discontinuations Due to AEs
Description: Subgroup analysis of on-treatment safety with non-cirrhosis vs cirrhosis, as measured by the frequency of SAEs, discontinuations due to AEs was conducted.
Time Frame: Up to post treatment week 4
Population: Subgroup analysis set included participants who received at least 1 dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | On-Treatment Safety of DCV 3DAA - Cirrhotic | On-Treatment Safety - Noncirrhotic
Number analyzed (Participants) | 23 | 146
Participants
  Serious AEs | 0 | 2
  AEs leading to Discontinuation | 1 | 3

12. Secondary Outcome: Number of Participants With/Without Cirrhosis as Measured by Selected Grade 3-4 Laboratory Abnormalities
Description: Subgroup analysis of on-treatment safety with non-cirrhosis vs cirrhosis, as measured by the selected Grade 3 - 4 laboratory abnormalities (including hematologic and liver function, based on DAIDS criteria) was conducted.
Time Frame: Up to post treatment week 4
Population: Subgroup analysis set included participants who received at least 1 dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | On-Treatment Safety of DCV 3DAA - Cirrhotic | On-Treatment Safety of DCV 3DAA - Noncirrhotic
Number analyzed (Participants) | 23 | 146
Participants
  Alanine Aminotransferase | 1 | 6
  Aspartate Aminotransferase | 1 | 4
  Lipase | 2 | 2
  Lymphocytes | 0 | 3
  Neutrophils | 1 | 1
  Hemoglobin | 0 | 1
  Platelets | 1 | 0
  International Normalized Ratio | 1 | 0
  Serum Glucose | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 12 Weeks within 30 days of discontinuation of dosing
Arm/Group | Treatment-Naive: DCV/ASV/BMS-791325 | Treatment-Experianced:
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/31
Serious Adverse Events (participants affected / at risk) | 2/138 | 0/31
Other Adverse Events (participants affected / at risk) | 62/138 | 20/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-Naive: DCV/ASV/BMS-791325 (N=138) | Treatment-Experianced: (N=31)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-Naive: DCV/ASV/BMS-791325 (N=138) | Treatment-Experianced: (N=31)
HEADACHE (Nervous system disorders) | 18 (19) | 4 (4)
DIZZINESS (Nervous system disorders) | 10 (11) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 10 (10) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 2 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 (14) | 3 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 11 (11) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (7) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 9 (10) | 3 (3)
FATIGUE (General disorders) | 6 (6) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication